CLINICAL TRIAL: NCT05203055
Title: A Multi-center, Open-label Study to Elucidate the Efficacy and Safety of Peginterferon Alpha-2b Therapy in the Initial Treatment of Chronic Hepatitis Patients With Normal ALT Level and Low Viremia
Brief Title: Peginterferon Alpha-2b Therapy in Chronic Hepatitis Patients With Normal ALT Level and Low Viremia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Peginterferon alpha-2b-HBV
Record Dates: First submitted 2021-12-18; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-12

CONDITIONS: Chronic Hepatitis B Patients With a Normal ALT Level and Low Viremia
MeSH Terms: interventions — peginterferon alfa-2b; Nucleotides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- monotherapy group (Experimental): Peginterferon alpha-2b injection is given subcutaneously at a dosage of 180μg/w for 48 consecutive weeks. Patients will stop the treatment whenever HBsAg is eliminated, and those without HBsAg elimination after 48 dosages will enter the group of best treatment. The patients will be followed up for another 24 weeks after treatment.
  Interventions: Drug: Peginterferon alpha-2b
- continuous combination therapy group (Experimental): Peginterferon alpha-2b injection is given subcutaneously at a dosage of 180μg/w for 48 consecutive weeks, plus continuous oral NA. Patients will stop the treatment whenever HBsAg is eliminated, and those without HBsAg elimination after 48 dosages will enter the group of best treatment. The patients will be followed up for another 24 weeks after treatment.
  Interventions: Drug: Peginterferon alpha-2b; Drug: Nucleotide Analog
- pulse combination therapy group (Experimental): Peginterferon alpha-2b injection is given subcutaneously at a dosage of 180μg/w for 8 consecutive weeks and cessation for 4 weeks,plus continuous oral NA. Patients will discontinue the treatment at any time if they are recovery, and those without HBsAg elimination after 48 dosages will enter the group of best treatment.The patients will be followed up for another 24 weeks after treatment.
  Interventions: Drug: Peginterferon alpha-2b; Drug: pulse peginterferon alpha-2b

INTERVENTIONS:
Drug: Peginterferon alpha-2b — 180μg/w
Drug: Nucleotide Analog — Etecavir 0.5mg qd or Tenofovir 300mg qd
  Arms: continuous combination therapy group
Drug: pulse peginterferon alpha-2b — 180μg/w for 8 consecutive weeks and cessation for 4 weeks
  Arms: pulse combination therapy group

SUMMARY:
To date, antiviral treatment is not recommended for chronic hepatitis B patients with a normal ALT level and low viremia. The strategy is to closely monitor the patients. However, evidence suggests that these group are at risk of gradual disease progression and development of hepatocellular carcinoma. Peginterferon eliminates the hepatitis B virus through immune regulation and induction of antiviral protein expression. For patients with low viral load, the clinical cure rate is potentially promising. In this study, we aim to investigate the efficacy and safety of peginterferon alpha-2b therapy in selected chronic hepatitis B patients with normal ALT level and low viremia. It is expected to obtain a satisfactory curative effect. Peginterferon is a marketed drug available in Chinese clinics with indications of anti-hepatitis B virus.

ELIGIBILITY:
Inclusion Criteria:

1. willing to receive the treatment and sign informed consent;
2. 18-60 years old (including 18 and 60), both gender;
3. HBsAg positive for at least 6 months and <1500IU/ml;
4. ALT≤1xULN and no elevated ALT has been detected in history;
5. HBV DNA detectable but<2000 IU/ml;
6. HBeAg negative ;

Exclusion Criteria:

1. For female participants: positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study. For male participants: intent to procreate 3 months before or after the intervention or unwillingness to use effective measures of the contraception ;
2. neuropsychiatric diseases, such as depression, anxiety, mania, schizophrenia, or a family history of mental illness (especially with a history of depression or depression tendency);
3. co-infection of HCV, EBV, other hepatotropic viruses , non-hepatotropic viruses;
4. alcoholic hepatitis, drug-induced hepatitis, autoimmune liver disease;
5. Patients with moderate to severe steatohepatitis;
6. possibility of liver cirrhosis that cannot be excluded
7. hepatocellular carcinoma or AFP level>30ng/ml;
8. Kidney diseases: acute and chronic nephritis, renal insufficiency, nephrotic syndrome, serum creatinine> 1 x ULN at the time of screening;
9. at screening, the neutrophil count is less than 1.5×10^9/L, and the platelet count is less than 90×10^9/L;
10. Serum phosphorus level <0.7 mmol/L;
11. Antinuclear antibody (ANA)>1:100;
12. Autoimmune diseases, including thyroiditis, psoriasis and systemic lupus erythematosus;
13. Endocrine system diseases, including thyroid diseases and diabetes mellitus;
14. Uncontrolled blood pressure: SBP>160 mmHg or DBP >100 mmHg at the time of enrollment;
15. Evidence of cardiovascular disease, existing congestive cardiac failure on physical exam and/or acute coronary syndrome in the past 6 months;
16. Severe retinopathy or other serious eye diseases;
17. Organic disease or dysfunction;
18. plan to receive an organ transplant or have already undergone an organ transplant;
19. received standardized treatment with interferon or NA products before .
20. allergic to interferon or pharmaceutical excipients, or meet any of the contraindications in the experimental drug instructions;
21. Participated in other interventional trials within 3 months before the screening or other conditions deemed unsuitable by the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with undetectable HBV DNA | week 24
HBsAg clearance rate | week 48
HBsAg conversion rate | week 48

SECONDARY OUTCOMES:
The percentage of patients with undetectable HBV DNA | week 24 and week 48
The HBsAg level | week 24 and week 48
The HBV pgRNA level | week 24 and week 48

CONTACTS AND LOCATIONS:
Locations (1):
- Fuzhou General Hospital, Xiamen Univ, Fuzhou, Fujian, China